CLINICAL TRIAL: NCT00581516
Title: Molecular Urine Tests for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Atreya Dash, MD, University of California, Irvine
Other Study IDs: 2006-5107
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PCA3
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Prostate cancer is the second leading cause of cancer related deaths among men in the United States.1 Although still controversial, there is growing evidence that early detection will reduce prostate cancer mortality. Currently the most useful biomarker to aid in early detection is measurement of serum prostate specific antigen (PSA) levels. Despite the value of PSA it has substantial limitations. To overcome the limitations of total PSA testing, there is emerging evidence demonstrating that relevant cancer biomarker can be detected in urine.

Patients who present to the urology clinic for a radical prostatectomy will be asked to enter this study. After obtaining informed consent, the following exam and specimen collection scheduled will be followed:

Visit 1 (pre-op):

Digital Rectal Exam (DRE) - Voided urine collection & serum collection

Visit 2 (time of prostatectomy):

Under anesthesia- catheterized urine collection and serum collection

Visit 3 (approximately 8 days post-prostatectomy):

Catheterized urine collection

Visit 4 (approximately 3 months post-prostatectomy):

Voided urine collection and serum collection

Some patients will not have the serum collection at visits 1, 2, and 4. The patients will be notified as to whether or not their blood will be drawn during the visits. Pre-operative Digital Rectal Exam, urinary catheterization and blood draws are part of standard of care in this patient population with localized prostate cancer. The catheter will be inserted during the time of surgery preparation in the operating room and removed during the post operative clinic appointment.

ELIGIBILITY:
Inclusion Criteria:

* Those scheduled to undergo radical prostatectomy for the treatment of prostate cancer.

Exclusion Criteria:

* minors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 male subjects who have clinically localized prostate cancer and are scheduled to undergo a radical prostatectomy are anticipated in this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atreya Dash, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States